CLINICAL TRIAL: NCT00368745
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Pregabalin in Subjects With Generalized Anxiety Disorder (GAD) Switching From Benzodiazepine Therapy.
Brief Title: Efficacy and Safety of Pregabalin vs Placebo for Generalized Anxiety Disorder (GAD) Symptoms in Subjects Discontinuing Benzodiazepine Treatment and Remaining 6 Weeks on Study Medication, Free From Benzodiazepine Use.
Acronym: GAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081092
Record Dates: First submitted 2006-08-23; First posted 2006-08-25 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2009-11

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin treatment for GAD during 6 week taper/discontinuation from alprazolam treatment; followed by 6 weeks pregabalin treatment 'alprazolam free'.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo treatment of GAD during 6 week taper/discontinuation of alprazolam treatment followed by 6 weeks continuation of placebo treatment 'alprazolam free'.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — GAD subjects on stable dose of alprazolam will be randomized to double-blind pregabalin at starting dose of 75mg twice daily. Weekly assessments of tolerability, need for rescue medication, anxiety/withdrawal symptoms will guide flexible dose titration of pregabalin at dose range between 75 and 300mg twice daily. Subjects successful in discontinuation of alprazolam while treated with pregabalin will continue to be maintained on pregabalin for 6 weeks and assessed weekly for ability to remain in the study.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — GAD subjects on stable dose of alprazolam will be randomized to double-blind placebo matching assessments and study medication titration as detailed under the pregabalin arm description. Subjects successful in discontinuation of alprazolam while treated with placebo will continue to be maintained on placebo for 6 weeks and assessed weekly for ability to remain in the study.
  Arms: Placebo

SUMMARY:
GAD subjects maintained on a stable dose of alprazolam for at least four weeks who meet eligibility criteria will be randomized to receive pregabalin vs matching placebo while simultaneously tapering off of alprazolam over 6 weeks. Subjects return weekly for assessment of safety/tolerability of pregabalin vs placebo as well as for assessment of anxiety and benzodiazepine withdrawal symptoms. Subjects successfully able to discontinue alprazolam, will continue 6 weeks of treatment with pregabalin vs placebo (free of benzodiazepine use). The efficacy and safety of pregabalin vs placebo for anxiety symptoms and ability to discontinue/remain free of alprazolam will be compared among pregabalin and placebo treated groups. Hypothesis is that a greater proportion of subjects will be successful in discontinuing and remaining free from benzodiazepines who were treated with pregabalin as compared to subjects treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* 18-65 years old
* male and female
* A primary lifetime diagnosis of DSM-IV-TR (2000) GAD (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition)

Exclusion Criteria:

* Pregnant or lactating women
* History of non-response to alprazolam, other benzodiazepines, gabapentin or pregabalin given for the treatment of anxiety as indicated by a (screening or baseline) Hamilton Anxiety Scale (HAM-A) score > 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Pfizer Investigational Site, San Pedro, Provincia de San José, Costa Rica
- Czechia (3):
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Praha-Bubenec
- France (5):
  - Pfizer Investigational Site, Paris, Cedex 12
  - Pfizer Investigational Site, Arcachon
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Élancourt
  - Pfizer Investigational Site, Nantes-Orvault
- Pfizer Investigational Site, Guatemala City, Guatemala
- Italy (2):
  - Pfizer Investigational Site, L’Aquila
  - Pfizer Investigational Site, Milan
- Mexico (3):
  - Pfizer Investigational Site, Tepic, Nayarit
  - Pfizer Investigational Site, Mexico City
  - Pfizer Investigational Site, San Luis Potosí City
- Spain (3):
  - Pfizer Investigational Site, Langreo, Principality of Asturias
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Zamora

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081092&StudyName=Efficacy%20and%20safety%20of%20pregabalin%20vs%20placebo%20for%20Generalized%20Anxiety%20disorder%20%28GAD%29%20symptoms%20in%20subjects%20discontinuing%20benzodiazepine%20tr

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, subjects were stabilized on a therapeutic dose of open-label alprazolam (minimum of 2 weeks) if they entered the study on a stable alprazolam dose or for up to 4 weeks if entered on a different benzodiazepine. Alprazolam dose range during 2-4 week stabilization phase was 1-4 milligrams (mg) by mouth (PO) twice a day (BID).
Groups:
- Pregabalin 75 mg to 300 mg PO BID: Pregabalin treatment following randomization to double-blind treatment: Baseline to Week 1: Pregabalin 75 mg PO BID (150 mg/day); Week 2: Pregabalin 150 mg PO BID (300 mg/day); Week 3 to Week 6 Pregabalin PO dosing ranged from 150 to 600 mg/day, given BID; during double-blind the alprazolam dose was tapered with a 25% reduction each week from baseline up to 6 weeks depending on the starting dose of alprazolam and toleration of dose reduction. Subjects successfully discontinued from alprazolam, continued for an additional 6 weeks of double-blind treatment with pregabalin at the same dose as during the double-blind taper.
- Placebo 75 mg to 300 mg PO BID: Placebo treatment following randomization to double-blind treatment: Baseline to Week 1: placebo 75 mg PO BID (150 mg/day); Week 2: placebo 150 mg PO BID (300 mg/day); Week 3 to Week 6 placebo PO dosing ranged from 150 to 600 mg/day, given BID; during double-blind the alprazolam dose was tapered with a 25% reduction each week from baseline up to 6 weeks depending on the starting dose of alprazolam and toleration of dose reduction. Subjects successfully discontinued from alprazolam, continued for an additional 6 weeks of double-blind treatment with placebo at the same dose as during the double-blind taper.
Period: Randomized to Double-blind Treatment
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Started | 57 | 51
Completed | 56 (One subject did not return following randomization; study drug not dispensed.) | 50 (One subject did not want to participate in study.)
Not Completed | 1 | 1
Period: Double-blind Treatment Period
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Started | 56 | 50
Completed | 30 | 19
Not Completed | 26 | 31
Not completed — Adverse Event | 6 | 6
Not completed — Lack of Efficacy | 7 | 16
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Other | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID | Total
Number analyzed (Participants) | 56 | 50 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.6) | 43.5 (11.3) | 41.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 76
  Male | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects at Endpoint (Post Alprazolam Free Week 6 or Last Observation Carried Forward [LOCF] Post Alprazolam Free Week 1) Who Are Benzodiazepine Free
Description: Number of subjects benzodiazepine free: < 2 doses rescue medication; negative urine benzodiazepine psychoactive toxicology assay (each visit Alprazolam Free phase); negative serum benzodiazepine alcohol assay (endpoint or LOCF).
Time Frame: Endpoint (Post Alprazolam Free Week 6 or LOCF Post Alprazolam Free Week 1)
Population: Intent to Treat (ITT) population: received at least 1 dose pregabalin or placebo. Primary outcome ITT = all treated subjects in alprazolam free phase. Endpoint = Post Alprazolam Free Week 6 or LOCF Post Alprazolam Free Week 1.
Measure: Number; unit: participants
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 37 | 27
participants | 20 | 10
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Primary objective: evaluate the efficacy of pregabalin in maintaining the benzodiazepine free state in subjects with prior stable alprazolam use; Test type: Superiority or Other; p = 0.2838, Cochran-Mantel-Haenszel — significance determined using 2-tailed significance level of 0.05; Cochran-Mantel-Haenszel (CMH) with country as a covariate

2. Secondary Outcome: Mean Change From Baseline in Hamilton Anxiety Scale (HAM-A) Scores
Description: HAM-A measures treatment-related changes in generalized anxiety symptoms; 14 item questionnaire scored 0 (not present) to 4 (very severe); lower score indicates less affected. Change from baseline: mean at observation minus mean at baseline.
Time Frame: Baseline, Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, and Endpoint (Alprazolam Free [AF] Week 6)
Population: ITT; subject has a baseline and at least 1 post-baseline measurement before week 13; endpoint = AF Week 6 or LOCF; (n) = number of subjects with data for analysis for pregabalin and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 46 | 41
scores on scale
  Alprazolam Taper (AT) Week 1 (n=46, 40) | -0.82 (0.66) | 0.67 (0.81)
  AT Week 2 (n=45, 37) | -1.72 (0.98) | 2.17 (1.15)
  AT Week 3 (n=33, 26) | -2.59 (0.99) | -0.21 (1.32)
  AT Week 4 (n=18, 11) | -1.47 (1.11) | 1.91 (1.82)
  AT Week 5 (n=8, 5) | -2.36 (2.19) | 2.86 (2.97)
  AT Week 6 (n=17, 9) | -1.26 (1.40) | 2.41 (2.11)
  Alprazolam Free (AF) Week 1 (n=39, 28) | -0.43 (0.90) | 2.40 (1.15)
  AF Week 2 (n=35, 24) | -2.15 (0.91) | -1.14 (1.19)
  AF Week 3 (n=31, 26) | -3.46 (0.92) | -2.47 (1.14)
  AF Week 4 (n=31, 19) | -3.58 (0.84) | -3.58 (1.14)
  AF Week 5 (n=27, 18) | -3.85 (0.87) | -3.34 (1.18)
  AF Week 6 (n=22, 15) | -5.62 (0.84) | -4.77 (1.05)
  Endpoint [LOCF] (n=46, 41) | -2.01 (1.13) | 2.77 (1.36)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Taper (AT) Week 1; Test type: Superiority or Other; p = 0.0709, ANCOVA — contrasts performed using Dunnett's Test; Least squares (LS) Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -1.48, 95% CI [-3.10 to 0.13], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 2; Test type: Superiority or Other; p = 0.0006, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -3.89, 95% CI [-6.04 to -1.74], Standard Error of Mean 1.08
Statistical Analysis 3: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 3; Test type: Superiority or Other; p = 0.0718, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -2.38, 95% CI [-4.98 to 0.22], Standard Error of Mean 1.30
Statistical Analysis 4: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 4; Test type: Superiority or Other; p = 0.0920, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -3.38, 95% CI [-7.37 to 0.60], Standard Error of Mean 1.92
Statistical Analysis 5: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT week 5; Test type: Superiority or Other; p = 0.1371, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -5.22, 95% CI [-12.67 to 2.23], Standard Error of Mean 3.04
Statistical Analysis 6: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 6; Test type: Superiority or Other; p = 0.0882, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -3.68, 95% CI [-7.96 to 0.61], Standard Error of Mean 2.04
Statistical Analysis 7: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Free (AF) Week 1; Test type: Superiority or Other; p = 0.0135, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -2.83, 95% CI [-5.05 to -0.61], Standard Error of Mean 1.11
Statistical Analysis 8: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 2; Test type: Superiority or Other; p = 0.3924, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -1.01, 95% CI [-3.38 to 1.35], Standard Error of Mean 1.18
Statistical Analysis 9: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 3; Test type: Superiority or Other; p = 0.3868, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -1.00, 95% CI [-3.29 to 1.30], Standard Error of Mean 1.14
Statistical Analysis 10: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 4; Test type: Superiority or Other; p = 0.9966, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = 0.00, 95% CI [-2.31 to 2.32], Standard Error of Mean 1.15
Statistical Analysis 11: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 5; Test type: Superiority or Other; p = 0.6873, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.51, 95% CI [-3.07 to 2.05], Standard Error of Mean 1.26
Statistical Analysis 12: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 6; Test type: Superiority or Other; p = 0.5337, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.85, 95% CI [-3.62 to 1.91], Standard Error of Mean 1.35
Statistical Analysis 13: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Endpoint [LOCF]; Test type: Superiority or Other; p = 0.0008, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -4.79, 95% CI [-7.51 to -2.07], Standard Error of Mean 1.37

3. Secondary Outcome: Number of Subjects With > = 6 Point Increase in Physician's Withdrawal Checklist (PWC) Scores
Description: PWC: 20 item physician rated interview (0 = not present; 3 = severe; score range: 0 to 60) measuring: signs of anxiolytic drug withdrawal and gastrointestinal (GI), mood, sleep, motor, somatic, perception and cognition symptoms. Data not analyzed: PWC not measured at baseline.
Time Frame: Baseline, Alprazolam Free Weeks 1 through 6, Endpoint (AF Week 6)
Population: ITT; data not analyzed: PWC not measured at baseline.
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Subjects With > = 5 New PWC Symptoms
Description: as for outcome 3
Time Frame: Baseline, Alprazolam Free Weeks 1 through 6, Endpoint (AF Week 6)
Population: ITT; data not analyzed: PWC not measured at baseline.
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 0 | 0

5. Post Hoc Outcome: Mean Scores Physician's Withdrawal Checklist (PWC)
Description: Mean scores at each visit for PWC: 20-item physician-rated interview measures presence of anxiolytic drug withdrawal-related signs and symptoms (gastrointestinal, mood, sleep, motor, somatic, perception, and cognition); range 0 (not present) to 3 (severe). Total score: 0 to 60; higher score = more affected. Mean scores entered as post-hoc analysis as Mean change from baseline in PWS scores not analyzed: PWS not measured at baseline.
Time Frame: Baseline, Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, Endpoint (AF Week 6 )
Population: ITT; (n) = number of subjects with data for analysis for pregabalin and placebo, respectively. Endpoint = AF Week 6 or LOCF. Refer to measure Mean Change From Baseline in Physician's Withdrawal Checklist (PWC) Scores.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 46 | 41
scores on scale
  Alprazolam Taper (AT) Week 1 (n=43, 40) | 6.32 (1.40) | 8.50 (1.45)
  AT Week 2 (n=44,37) | 6.37 (1.18) | 10.00 (1.34)
  AT Week 3 (n=33, 26) | 6.56 (1.40) | 9.41 (1.76)
  AT Week 4 (n=18, 11) | 5.63 (0.89) | 9.04 (1.37)
  AT Week 5 (n=7, 5) | 7.30 (1.52) | 9.58 (2.32)
  AT Week 6 (n=17, 9) | 6.82 (1.39) | 12.55 (2.07)
  Alprazolam Free (AF) Week 1 (n=39, 28) | 6.78 (1.15) | 10.70 (1.45)
  AF Week 2 (n=33, 24) | 4.71 (0.93) | 6.43 (1.19)
  AF Week 3 (n=30, 26) | 6.86 (0.85) | 7.16 (1.05)
  AF Week 4 (n=30, 19) | 7.43 (0.89) | 6.99 (1.17)
  AF Week 5 (n=27, 18) | 7.87 (0.76) | 8.25 (1.00)
  AF Week 6 (n=22, 15) | 2.40 (0.94) | 5.51 (1.16)
  Endpoint [LOCF] (n=46, 41) | 6.48 (1.23) | 10.28 (1.44)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Taper (AT) Week 1; Test type: Superiority or Other; p = 0.1220, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -2.18, 95% CI [-4.97 to 0.60], Standard Error of Mean 1.40
Statistical Analysis 2: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 2; Test type: Superiority or Other; p = 0.0053, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -3.63, 95% CI [-6.15 to -1.11], Standard Error of Mean 1.26
Statistical Analysis 3: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 3; Test type: Superiority or Other; p = 0.1048, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -2.85, 95% CI [-6.32 to 0.62], Standard Error of Mean 1.73
Statistical Analysis 4: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 4; Test type: Superiority or Other; p = 0.0357, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -3.41, 95% CI [-6.57 to -0.25], Standard Error of Mean 1.52
Statistical Analysis 5: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 5; Test type: Superiority or Other; p = 0.4263, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -2.28, 95% CI [-8.82 to 4.26], Standard Error of Mean 2.67
Statistical Analysis 6: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 6; Test type: Superiority or Other; p = 0.0104, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -5.73, 95% CI [-9.96 to -1.51], Standard Error of Mean 2.02
Statistical Analysis 7: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Free (AF) Week 1; Test type: Superiority or Other; p = 0.0069, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -3.92, 95% CI [-6.73 to -1.12], Standard Error of Mean 1.40
Statistical Analysis 8: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 2; Test type: Superiority or Other; p = 0.2185, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -1.71, 95% CI [-4.47 to 1.05], Standard Error of Mean 1.37
Statistical Analysis 9: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 3; Test type: Superiority or Other; p = 0.7832, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.29, 95% CI [-2.41 to 1.83], Standard Error of Mean 1.06
Statistical Analysis 10: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 4; Test type: Superiority or Other; p = 0.7062, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = 0.44, 95% CI [-1.90 to 2.79], Standard Error of Mean 1.16
Statistical Analysis 11: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 5; Test type: Superiority or Other; p = 0.7161, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.38, 95% CI [-2.49 to 1.73], Standard Error of Mean 1.04
Statistical Analysis 12: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 6; Test type: Superiority or Other; p = 0.0376, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -3.11, 95% CI [-6.03 to -0.19], Standard Error of Mean 1.43
Statistical Analysis 13: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Endpoint [LOCF]; Test type: Superiority or Other; p = 0.0122, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -3.80, 95% CI [-6.74 to -0.85], Standard Error of Mean 1.48

6. Secondary Outcome: Mean Change From Baseline in Physician's Withdrawal Checklist (PWC) Scores
Description: PWC: 20 item physician rated interview (0 = not present; 3 = severe; score range: 0 to 60) measuring: signs of anxiolytic drug withdrawal and gastrointestinal (GI), mood, sleep, motor, somatic, perception and cognition symptoms. Change from baseline not analyzed as PWC was not measured at baseline. Mean PWS scores presented in Post-hoc outcome measure Mean PWS scores.
Time Frame: Baseline, Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, Endpoint (AF Week 6)
Population: ITT; Change from baseline not analyzed as PWC was not measured at baseline. Mean PWS scores presented in Post-hoc outcome measure Mean PWS scores.
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale Scores.
Description: CGI-S: 7-point scale to assess global change in subject condition compared to baseline; range 1 (no evidence of illness) to 7 (among the most severely ill); higher score = more affected. Change from baseline: mean at observation minus mean at baseline.
Time Frame: Baseline, Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, and Endpoint (AF Week 6 )
Population: ITT; subject has a baseline and at least 1 post-baseline endpoint measurement; endpoint = AF Week 6 or LOCF; (n) = number of subjects with data for analysis for pregabalin and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 45 | 41
scores on scale
  Alprazolam Taper (AT) Week 1 (n=45, 40) | -0.23 (0.13) | 0.22 (0.15)
  AT Week 2 (n=44, 37) | -0.33 (0.17) | 0.41 (0.19)
  AT Week 3 (n=32, 27) | -0.60 (0.20) | -0.10 (0.26)
  AT Week 4 (n=17, 11) | -0.41 (0.21) | -0.04 (0.32)
  AT Week 5 (n=7, 5) | -0.77 (0.27) | -0.05 (0.40)
  AT Week 6 (n=16, 9) | -0.63 (0.32) | 0.08 (0.43)
  Alprazolam Free (AF) Week 1 (n=38, 28) | -0.46 (0.17) | 0.23 (0.21)
  AF Week 2 (n=34, 24) | -0.98 (0.20) | -0.48 (0.26)
  AF Week 3 (n=30, 26) | -0.88 (0.22) | -0.32 (0.27)
  AF Week 4 (n=30, 19) | -0.87 (0.18) | -0.84 (0.25)
  AF Week 5 (n=26, 18) | -0.82 (0.19) | -0.75 (0.26)
  AF Week 6 (n=21, 15) | -1.33 (0.20) | -1.02 (0.25)
  Endpoint [LOCF] (n=45, 41) | -0.45 (0.21) | 0.31 (0.24)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Taper (AT) Week 1; Test type: Superiority or Other; p = 0.0052, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.45, 95% CI [-0.76 to -0.14], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 2; Test type: Superiority or Other; p = 0.0001, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.74, 95% CI [-1.11 to -0.38], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 3; Test type: Superiority or Other; p = 0.0528, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.50, 95% CI [-1.00 to 0.01], Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 4; Test type: Superiority or Other; p = 0.3085, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.37, 95% CI [-1.11 to 0.37], Standard Error of Mean 0.35
Statistical Analysis 5: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 5; Test type: Superiority or Other; p = 0.1807, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.72, 95% CI [-1.92 to 0.47], Standard Error of Mean 0.47
Statistical Analysis 6: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 6; Test type: Superiority or Other; p = 0.1074, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.71, 95% CI [-1.58 to 0.17], Standard Error of Mean 0.42
Statistical Analysis 7: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Free (AF) Week 1; Test type: Superiority or Other; p = 0.0013, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.69, 95% CI [-1.10 to -0.28], Standard Error of Mean 0.20
Statistical Analysis 8: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 2; Test type: Superiority or Other; p = 0.0503, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.50, 95% CI [-0.99 to 0.00], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 3; Test type: Superiority or Other; p = 0.0364, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.56, 95% CI [-1.09 to -0.04], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 4; Test type: Superiority or Other; p = 0.9140, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.03, 95% CI [-0.51 to 0.46], Standard Error of Mean 0.24
Statistical Analysis 11: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 5; Test type: Superiority or Other; p = 0.7789, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.08, 95% CI [-0.62 to 0.47], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 6; Test type: Superiority or Other; p = 0.3189, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.32, 95% CI [-0.95 to 0.32], Standard Error of Mean 0.31
Statistical Analysis 13: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Endpoint [LOCF]; Test type: Superiority or Other; p = 0.0031, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as covariate; Mean Difference (Final Values) = -0.76, 95% CI [-1.26 to -0.27], Standard Error of Mean 0.25

8. Secondary Outcome: Mean Scores for Clinical Global Impression-Improvement (CGI-I) Scale
Description: CGI-I: 7-point scale to assess global change in subject condition compared to baseline; range 1 (very much improved) to 7 (very much worse); higher score = more affected.
Time Frame: Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, and Endpoint (AF Week 6 )
Population: ITT; subject has a baseline and endpoint measurement; endpoint = AF Week 6 or LOCF; (n) = number of subjects with data for analysis for pregabalin and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 46 | 41
scores on scale
  Alprazolam Taper (AT) Week 1 (n=46, 39) | 3.52 (0.20) | 3.90 (0.24)
  AT Week 2 (n=45, 37) | 3.17 (0.27) | 3.98 (0.31)
  AT Week 3 (n=33, 27) | 2.88 (0.31) | 3.47 (0.39)
  AT Week 4 (n=18, 11) | 3.09 (0.35) | 3.01 (0.54)
  AT Week 5 (n=8, 5) | 2.63 (0.30) | 3.44 (0.47)
  AT Week 6 (n=17, 9) | 3.00 (0.31) | 3.86 (0.46)
  Alprazolam Free (AF) Week 1 (n=39, 28) | 2.93 (0.28) | 3.90 (0.36)
  AF Week 2 (n=35, 24) | 2.39 (0.28) | 3.27 (0.35)
  AF Week 3 (n=30, 26) | 2.15 (0.28) | 2.93 (0.35)
  AF Week 4 (n=31, 19) | 2.20 (0.29) | 2.46 (0.39)
  AF Week 5 (n=27, 18) | 2.29 (0.32) | 2.77 (0.42)
  AF Week 6 (n=22, 15) | 1.52 (0.28) | 2.18 (0.34)
  Endpoint [LOCF] (n= 46, 41) | 2.57 (0.30) | 3.52 (0.35)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Taper (AT) Week 1; Test type: Superiority or Other; p = 0.1260, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.37, 95% CI [-0.86 to 0.11], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 2; Test type: Superiority or Other; p = 0.0074, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.81, 95% CI [-1.40 to -0.22], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 3; Test type: Superiority or Other; p = 0.1250, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.59, 95% CI [-1.35 to 0.17], Standard Error of Mean 0.38
Statistical Analysis 4: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 4; Test type: Superiority or Other; p = 0.8991, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = 0.08, 95% CI [-1.17 to 1.32], Standard Error of Mean 0.60
Statistical Analysis 5: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 5; Test type: Superiority or Other; p = 0.1747, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.81, 95% CI [-2.07 to 0.46], Standard Error of Mean 0.53
Statistical Analysis 6: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 6; Test type: Superiority or Other; p = 0.0744, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.85, 95% CI [-1.79 to 0.09], Standard Error of Mean 0.45
Statistical Analysis 7: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Free (AF) Week 1; Test type: Superiority or Other; p = 0.0063, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.98, 95% CI [-1.67 to -0.29], Standard Error of Mean 0.35
Statistical Analysis 8: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 2; Test type: Superiority or Other; p = 0.0140, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.87, 95% CI [-1.56 to -0.18], Standard Error of Mean 0.34
Statistical Analysis 9: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 3; Test type: Superiority or Other; p = 0.0267, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.78, 95% CI [-1.46 to -0.09], Standard Error of Mean 0.34
Statistical Analysis 10: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 4; Test type: Superiority or Other; p = 0.5104, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.26, 95% CI [-1.03 to 0.52], Standard Error of Mean 0.38
Statistical Analysis 11: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 5; Test type: Superiority or Other; p = 0.2702, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.48, 95% CI [-1.35 to 0.39], Standard Error of Mean 0.43
Statistical Analysis 12: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 6; Test type: Superiority or Other; p = 0.1241, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.66, 95% CI [-1.52 to 0.19], Standard Error of Mean 0.42
Statistical Analysis 13: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Endpoint [LOCF]; Test type: Superiority or Other; p = 0.0109, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.95, 95% CI [-1.67 to -0.22], Standard Error of Mean 0.36

9. Secondary Outcome: Mean Scores for Patient Global Impression-Improvement (PGI-I)
Description: PGI-I: subject rated 7-point scale measures change in overall status; range 1 (very much improved) to 7 (very much worse).
Time Frame: Alprazolam Taper Weeks 1 through 6, Alprazolam Free Weeks 1 through 6, and Endpoint (AF Week 6 )
Population: ITT; endpoint = AF Week 6 or LOCF; (n) = number of subjects with data for analysis for pregabalin and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 46 | 41
scores on scale
  Alprazolam Taper (AT) Week 1 (n=46, 40) | 3.16 (0.23) | 3.82 (0.27)
  AT Week 2 (n= 45, 37) | 3.13 (0.32) | 4.03 (0.36)
  AT Week 3 (n=33, 26) | 2.93 (0.28) | 3.31 (0.35)
  AT Week 4 (n=18, 11) | 3.12 (0.34) | 2.98 (0.52)
  AT Week 5 (n=8, 5) | 2.91 (0.37) | 3.75 (0.58)
  AT Week 6 (n=17, 9) | 2.93 (0.42) | 3.38 (0.63)
  Alprazolam Free (AF) Week 1 (n=39, 28) | 2.95 (0.26) | 3.45 (0.33)
  AF Week 2 (n=35, 24) | 2.34 (0.27) | 2.94 (0.34)
  AF Week 3 (n=31, 26) | 2.28 (0.28) | 2.92 (0.35)
  AF Week 4 (n=30, 19) | 2.43 (0.29) | 2.73 (0.38)
  AF Week 5 (n=27, 18) | 2.32 (0.31) | 2.70 (0.41)
  AF Week 6 (n=22, 14) | 1.53 (0.27) | 2.48 (0.35)
  Endpoint [LOCF] (n=46, 41) | 2.71 (0.32) | 3.74 (0.38)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Taper (AT) Week 1; Test type: Superiority or Other; p = 0.0226, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.66, 95% CI [-1.22 to -0.09], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 2; Test type: Superiority or Other; p = 0.0099, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.90, 95% CI [-1.58 to -0.22], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 3; Test type: Superiority or Other; p = 0.2827, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.38, 95% CI [-1.07 to 0.32], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 4; Test type: Superiority or Other; p = 0.8232, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = 0.13, 95% CI [-1.07 to 1.34], Standard Error of Mean 0.58
Statistical Analysis 5: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 5; Test type: Superiority or Other; p = 0.2409, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.85, 95% CI [-2.41 to 0.72], Standard Error of Mean 0.66
Statistical Analysis 6: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AT Week 6; Test type: Superiority or Other; p = 0.4760, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.45, 95% CI [-1.73 to 0.84], Standard Error of Mean 0.61
Statistical Analysis 7: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Alprazolam Free (AF) Week 1; Test type: Superiority or Other; p = 0.1252, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.50, 95% CI [-1.14 to 0.14], Standard Error of Mean 0.32
Statistical Analysis 8: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 2; Test type: Superiority or Other; p = 0.0717, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.60, 95% CI [-1.26 to 0.06], Standard Error of Mean 0.33
Statistical Analysis 9: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 3; Test type: Superiority or Other; p = 0.0707, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.64, 95% CI [-1.33 to 0.06], Standard Error of Mean 0.35
Statistical Analysis 10: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 4; Test type: Superiority or Other; p = 0.4341, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.30, 95% CI [-1.08 to 0.47], Standard Error of Mean 0.39
Statistical Analysis 11: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 5; Test type: Superiority or Other; p = 0.3700, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.38, 95% CI [-1.23 to 0.47], Standard Error of Mean 0.42
Statistical Analysis 12: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; AF Week 6; Test type: Superiority or Other; p = 0.0328, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -0.96, 95% CI [-1.83 to -0.08], Standard Error of Mean 0.43
Statistical Analysis 13: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Endpoint [LOCF]; Test type: Superiority or Other; p = 0.0096, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country as covariate; Mean Difference (Final Values) = -1.03, 95% CI [-1.80 to -0.26], Standard Error of Mean 0.39

10. Secondary Outcome: Mean Change From Baseline in Digit Symbol Substitution Test (DSST) Scores
Description: DSST: subject-rated; evaluates aspects of cognition (includes attending to directions, processing speed, sustained attention, visual-motor integration, learning and psychomotor speed). Subject matches symbol (1 to 9) with corresponding number key (1 to 9); number of correct symbol-number pairs completed by subject over a 90-second test period determines DSST score. Change: mean at observation minus mean at baseline. Data summarized as change from baseline to endpoint.
Time Frame: Baseline, Endpoint (AF Week 6 )
Population: ITT; subject has baseline and endpoint (final visit) measurement; endpoint = AF Week 6 or LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 33 | 29
scores on scale | 13.10 (2.64) | 13.47 (2.95)
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Test type: Superiority or Other; p = 0.8897, ANCOVA — contrasts performed using Dunnett's Test; LS Means from the ANCOVA model with treatment as the main effect and country and baseline as the covariate; Mean Difference (Final Values) = -0.37, 95% CI [-5.74 to 4.99], Standard Error of Mean 2.68

11. Secondary Outcome: Time to Discontinuation
Description: The 25th percentile estimate of time until discontinuation is based on Kaplan-Meier estimates. Event day is the study day when the subject discontinued from study.
Time Frame: Baseline, Week 13 (Final Visit/Early Termination)
Population: ITT; Week 13 (Final Visit/Early Termination) or LOCF.
Measure: Number; unit: days
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 19 | 24
days | 51 | 33
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Test type: Superiority or Other; p = 0.0626, Log Rank — p-value is from the log-rank statistic from the tests for equality over treatment as strata and country used as covariate

12. Secondary Outcome: Time to First Use of Rescue Medication
Description: The 25th percentile estimate of time until first use of rescue medication is based on Kaplan-Meier estimates. Event day is the study day when the subject first used rescue medication. Rescue medication: packet with 2 doses alprazolam to take only in the event subject experiences severe symptoms of benzodiazepine withdrawal or rebound anxiety.
Time Frame: Baseline, Week 13 (Final Visit/Early Termination)
Population: ITT; Week 13 (Final Visit/Early Termination) or LOCF
Measure: Number; unit: days
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 11 | 17
days | 63 | 30
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Test type: Superiority or Other; p = 0.0148, Log Rank — [p-value comment as in outcome 11, analysis 1]

13. Secondary Outcome: Number of Subjects in Relapse Free State at 6-week Benzodiazepine-free Endpoint (Alprazolam Free Week 6)
Description: Number of subjects benzodiazepine free: < 2 doses rescue medication; negative urine toxicology assay (each visit Alprazolam Free phase), negative urine alcohol assay (Alprazolam Free Week 6 = endpoint or LOCF). Relapse: > = 2 intakes rescue medication, positive urine and /or alcohol assays, unable to tolerate alprazolam taper, or discontinuation.
Time Frame: Alprazolam Free Week 6
Population: ITT; endpoint = AF Week 6 or LOCF.
Measure: Number; unit: participants
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Number analyzed (Participants) | 22 | 15
participants | 21 | 12
Statistical Analysis 1: Comparison: Pregabalin 75 mg to 300 mg PO BID vs Placebo 75 mg to 300 mg PO BID; Test type: Superiority or Other; p = 0.1159, Cochran-Mantel-Haenszel — p-value is obtained using Cochran-Mantel-Haenszel option

ADVERSE EVENTS:
Arm/Group | Pregabalin 75 mg to 300 mg PO BID | Placebo 75 mg to 300 mg PO BID
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/50
Other Adverse Events (participants affected / at risk) | 33/56 | 29/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 75 mg to 300 mg PO BID (N=56) | Placebo 75 mg to 300 mg PO BID (N=50)
Hyperacusis (Ear and labyrinth disorders) | 3 | 1
Vision blurred (Eye disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 5 | 7
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 3 | 5
Fatigue (General disorders) | 2 | 3
Irritability (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 12 | 3
Headache (Nervous system disorders) | 7 | 13
Paraesthesia (Nervous system disorders) | 6 | 0
Somnolence (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 11 | 10
Insomnia (Psychiatric disorders) | 4 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.